CLINICAL TRIAL: NCT04816682
Title: Does Silymarin Mitigate Clinical Course of COVID-19 in Patients Admitted to an Internal Medicine Ward With Elevated Liver Enzymes?
Brief Title: Silymarin in COVID-19 Patients Admitted to Hospital With Elevated Liver Enzymes
Acronym: SILCOVINT-21
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: F.D. Roosevelt Teaching Hospital with Policlinic Banska Bystrica (Other)
Responsible Party: Principal Investigator, Ľubomír Skladaný MD, PhD, Head, Department of Internal Medicine and HEGITO Liver Unit, Principal Investigator, F.D. Roosevelt Teaching Hospital with Policlinic Banska Bystrica
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SIL-COVINT-21
Record Dates: First submitted 2021-03-19; First posted 2021-03-25 (Actual); Last update posted 2022-08-03 (Actual); Status verified 2022-08

CONDITIONS: Covid19; Liver Diseases
Keywords: COVID-19; In-hospital mortality; Internal medicine
MeSH Terms: conditions — COVID-19; Liver Diseases | interventions — Silymarin; Silybin

STUDY DESIGN:
Intervention Model Description: Prospective open label study using historical cohort for propensity-match analysis
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LAGOSA ARM (Active Comparator): Consecutively admitted patients will be allocated silymarin tablets (150 mg each) T.I.D. 3-2-2
  Interventions: Drug: Silymarin
- Control arm (No Intervention): Consecutive patients with the same inclusion/exclusion criteria as in active arm, hospitalised at the same department before the initiation of the study (historical controls)

INTERVENTIONS:
Drug: Silymarin — Silymarine tablets will be provided irrespective of meal by a registered nurse T.I.D
  Other Names: LAGOSA
  Arms: LAGOSA ARM

SUMMARY:
Of patients admitted to an internal medicine ward with internistic diagnosis/es together with COVID-19, substantial proportion has elevated liver enzymes. silymarin / silibinin (milk thistle extract) has been approved as an add-on therapy in various acute and chronic liver diseases; moreover, there is evidence to suggest that it's dual effect (anti-viral and immune-modulatory) might be of benefit in patients infected with SARS-CoV-2. As there is no effective/approved pharmacotherapy for COVID-19, a pilot study with Silymarine in hospitalised patients has been undertaken

DETAILED DESCRIPTION:
According to the Bosch-Barrera et al. paper of 2021, silibinin in a daily dose of more than 1000 mg could improve clinical course of COVID-19 by its dual action: 1.direct inhibition of SARS-CoV-2 replication as well as 2.modulation of innate immune response - 2a. its initial (hyper)inflammation as well as 2b. later reparative phase, respectively.

Moreover, the drug is known for its safety and has been approved and widely used in the region for liver diseases. Therefore, the investigation was set out to determine the efficacy of silymarin (compound closely related to Silibinin which is available in the region) in improving the outcome of a liver disease and of COVID-19, respectively.

ELIGIBILITY:
Inclusion Criteria:

* consecutive, adult, admitted to an internal medicine ward with internistic diagnosis, together with COVID-19, and elevated liver enzymes (any of AST, ALT, GGT, ALP), provided written informed consent

Exclusion Criteria:

* too sick - terminal illness (no potential for recovery); critical condition on admission requiring immediate tracheal intubation; or any extra-pulmonary organ failure; completely vaccinated against COVID19.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-03-17 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
Improvement in the COVID-19 stage of at least 1 point | During the hospital stay - up to around 21 days
  Evolution of COVID-19 will be recorded according to a WHO criteria and reported as worsening (including death) / no change / improvement
Improvement in the activity of aminotranspherases | During the hospital stay - up to around 21 days
  Change in the level of ALT

SECONDARY OUTCOMES:
Improvement in the diabetes control | During the hospital stay - up to around 21 days
  Change in the glycemia
Improvement in the blood inflammatory markers | During the hospital stay - up to around 21 days
  Change in C-reactive protein levels
Improvement in the dyspnea | During the hospital stay - up to around 21 days
  Improvement of at least one point in the NYHA classification
Improvement in the acute kidney injury | During the hospital stay - up to around 21 days
  Any improvement in the serum creatinine level
Improvement in the blood inflammatory markers | During the hospital stay - up to around 21 days
  Improvement in the interleukin - 6 level

CONTACTS AND LOCATIONS:
Overall Officials: Lubomir SKLADANY, MD, PhD, Principal Investigator — Study Principal Investigator F.D.Roosevelt Teaching Hospital, Banska Bystrica, Slovakia
Locations (2):
- Slovakia (2):
  - F.D.Roosevelt Teaching Hospital, Banská Bystrica
  - University Hospital Bratislava, Bratislava

IPD SHARING:
Plan to Share IPD: Yes
Complete dataset will be shared on request under GDPR rules
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Dataset / protocol / ICF will be open for audit anytime Dataset will be shared after completion of upload
Access Criteria: Journal editors Investigators - by the hypothesis testable on the dataset Auditing authority
URL: http://www.fnspfdr.sk

REFERENCES:
- [Result] Bosch-Barrera J, Martin-Castillo B, Buxo M, Brunet J, Encinar JA, Menendez JA. Silibinin and SARS-CoV-2: Dual Targeting of Host Cytokine Storm and Virus Replication Machinery for Clinical Management of COVID-19 Patients. J Clin Med. 2020 Jun 7;9(6):1770. doi: 10.3390/jcm9061770. PMID 32517353